CLINICAL TRIAL: NCT03613467
Title: Vedio-assisted Thoracoscopic Lobectomy vs Open Lobectomy for Patients With Surgically Resectable Pathologic N2 NSCLC
Brief Title: Is Video-assisted Thoracoscopic Lobectomy a Clinical Alternative for Surgically Resectable Pathologic N2 NSCLC Patients
Status: Completed | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Collaborators: LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, lixiaofei, Professor, Tang-Du Hospital
Other Study IDs: W-TONG06
Record Dates: First submitted 2018-07-16; First posted 2018-08-03 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Vedio-assisted thoracoscopic lobectomy; Thoracotomy lobectomy; Real-world evidences;; pN2 NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VATS lobectomy: Pathologic N2 NSCLC patients who received lobectomy by video-assisted thoracoscopic surgery
  Interventions: Procedure: VATS lobectomy
- Thoracotomy lobectomy: Pathologic N2 NSCLC patients who received lobectomy by thoracotomy
  Interventions: Procedure: Thoracotomy lobectomy

INTERVENTIONS:
Procedure: VATS lobectomy — Patients who received lobectomy by video-assisted thoracoscopic surgery
  Groups: VATS lobectomy
Procedure: Thoracotomy lobectomy — Patients who received lobectomy by thoracotomy
  Groups: Thoracotomy lobectomy

SUMMARY:
The study was designed to compare the safety and effectiveness of vedio-assisted thoracoscopic lobectomy with open lobectomy for patients with surgically resectable pathologic N2 non-small cell lung cancer

DETAILED DESCRIPTION:
The is a multi-center retrospective study. Patients with pathologic N2 NSCLC who underwent VATS or open lobectomy between 2014 and 2017 were included into this study. Clinical data on patient demographic, clinical characteristics, treatment and clinical outcomes will be collected to evaluate the safety and effectiveness of video-assisted thoracoscopic lobectomy for pathologic N2 NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age > 18 years old;
* Patients with pathologically diagnosed non-small cell lung cancer;
* Patients underwent lobectomy by either VATS or thoracotomy between 2014 and 2017;
* Patients who received lymphadenectomy for all accessible lymph nodes;
* Patients with N2 lymph nodes (+) after surgeries;

Exclusion Criteria:

* Patients with second primary tumors or multiple primary tumors;
* Patients who received chest surgeries before hospitalization;
* Patients with superior pulmonary sulcus tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically diagnosed N2 non-small cell lung cancer who received VATS or thoracotomy lobectomy between 2014 and 2017
Sampling Method: Non-Probability Sample
Enrollment: 2145 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2014-2018
  Overall survival

SECONDARY OUTCOMES:
Duration of hospital stay [Perioperative outcomes] | 2014-2017
  Duration of hospital stay [Perioperative outcomes]
Postoperative 30 and 90 days [Perioperative outcomes] | 2014-2017
  Postoperative 30 and 90 days [Perioperative outcomes]
Drainage time [Perioperative outcomes] | 2014-2017
  Drainage time [Perioperative outcomes]
Intraoperative blood loss [Perioperative outcomes] | 2014-2017
  Intraoperative blood loss [Perioperative outcomes]
Postoperative complications [Perioperative outcomes] | 2014-2017
  Postoperative complications [Perioperative outcomes]

OTHER OUTCOMES:
Overall survivals in the subgroups stratified by T staging | 2014-2018
  Overall survivals in the subgroups stratified by T staging
Overall survivals in the subgroups stratified by neoadjuvant therapy | 2014-2018
  Overall survivals in the subgroups stratified by neoadjuvant therapy
Overall survivals in the subgroups stratified by number of lymph node station involved | 2014-2018
  Overall survivals in the subgroups stratified by number of lymph node station involved
Impact factors for overall survival | 2014-2018
  Impact factors for overall survival
Impact factors for postoperative mortality within 30/90 days | 2014-2017
  Impact factors for postoperative mortality within 30/90 days
Propensity score matching analysis of overall survival | 2014-2018
  Propensity score matching analysis of overall survival
Propensity score matching analysis of perioperative outcomes | 2014-2018
  Propensity score matching analysis of perioperative outcomes
Propensity score matching analysis of impact factors for overall survival | 2014-2018
  Propensity score matching analysis of impact factors for overall survival
Propensity score matching analysis of impact factors for postoperative mortality within 30/90 days | 2014-2018
  Propensity score matching analysis of impact factors for postoperative mortality within 30/90 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofei Li, PhD, Principal Investigator — Tang-Du Hospital
Locations (10):
- China (10):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - China PLA General Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Huazhong Technology Hospital, Wuhan, Hubei
  - Jiangsu cancer hospital, Nanjing, Jiangsu
  - Xi'an Tangdu Hospital, Xi'an, Shaanxi
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Huaxi Hospital Affiliated to Sichuan University, Chengdu, Sichuan
  - Tianjin Chest Hospital, Tianjin, Tianjin Municipality
  - First Hospital Affiliated to Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No